CLINICAL TRIAL: NCT05893875
Title: Exploring the Changes of Inflammatory Factors in Joint Fluid of Patients With Sports Injury for 1-year Postoperative Rehabilitation and Clinical Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-553-01
Record Dates: First submitted 2023-05-27; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to use a prospective study design method to continuously collect immune cell and inflammatory factor data of 5ml peripheral blood and 10ml joint fluid from 200 patients who met the inclusion and exclusion criteria in our department from January 2020 to January 2022. The aim is to analyze the impact of changes in inflammatory factors before and after surgery on postoperative recovery.

DETAILED DESCRIPTION:
This study intends to use a retrospective study design method to continuously collect immune cell and inflammatory factor data of 5ml peripheral blood and 10ml joint fluid from 200 patients who met the inclusion and exclusion criteria in our department starting from January 2021. The aim is to analyze the impact of changes in inflammatory factors before and after surgery on postoperative recovery. The indicators of postoperative rehabilitation for patients were objectively evaluated using three scales: Lysholm scale, VAS scale, and Tegner scale. Among them, the Lysholm scale mainly evaluates the postoperative recovery of knee joint function in patients, with values ranging from 0 to 100. The higher the value, the better the recovery; The VAS scale mainly evaluates the postoperative pain score of patients, with values ranging from 0 to 10. The higher the value, the more severe the pain; The Tegner scale is also mainly used to evaluate the postoperative recovery of knee joint function in patients, with values ranging from 0 to 10. The higher the value, the better the recovery.

ELIGIBILITY:
Inclusion Criteria:

* Those with healthy diet and regular exercise habits;
* Sports injury patients(Satisfy one of the following conditions): Anterior cruciate ligament injury or meniscus injury

Exclusion Criteria:

* Existence of underlying diseases related to the immune system;
* Trauma leading to knee joint fracture;
* Blood pressure, heart rate, vital capacity, muscle tension and other indicators are obviously abnormal;
* Significant abnormalities in blood routine, infection indicators, heart, lung, liver, and kidney function tests, insufficient compensatory function of important organs, or severe systemic diseases;
* Patients with neurological or psychiatric disorders, pregnant women, or a history of related illnesses combined with severe organic diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who underwent anterior cruciate ligament reconstruction surgery at the Sports Medicine Department of Sun Yat sen Memorial Hospital and required joint effusion extraction due to postoperative treatment
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score for pain (VAS) | Change from 2 weeks, 1 month, 3 months, 6 months, and 1 Year after ACLR operation
  The VAS scale mainly evaluates the postoperative pain score of patients, with values ranging from 0 to 10. The higher the value, the more severe the pain;
Lysholm score | Change from 6 months and 1 Year after ACLR operation
  The Lysholm scale mainly evaluates the postoperative recovery of knee joint function in patients, with values ranging from 0 to 100. The higher the value, the better the recovery;
Tegner sacle | Change from 6 months and 1 Year after ACLR operation
  The Tegner scale is also mainly used to evaluate the postoperative recovery of knee joint function in patients, with values ranging from 0 to 10. The higher the value, the better the recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yatsen Memorial Hospital, Guangzhou, Guangdong, China